CLINICAL TRIAL: NCT05202639
Title: Decision-making Regarding the Possibility of Medical Termination of Pregnancy on Two Multidisciplinary Prenatal Diagnosis Centers of Maternities Level 3 in Lyon in 2019
Brief Title: Decision-making Regarding the Possibility of Medical Termination of Pregnancy
Acronym: DEFIMEG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0580
Record Dates: First submitted 2021-12-14; First posted 2022-01-21 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Medical Termination of Pregnancy
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Continuation of pregnancy: The parents who have chosen to continue pregnancy will be asked to complete a questionnaire.
  Interventions: Other: Questionnaire
- Medical termination of pregnancy: The parents who have chosen to terminate pregnancy will be asked to complete a questionnaire.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire will be sent by e-mail to the mother and to the father separately. A return of the completed questionnaire is expected within 6 weeks via a secure internal platform pertained to the HCL ("Hospices Civils de Lyon").
  The aim of this questionnaire is to identify the factors associated with the continuation or not of pregnancy after diagnosis of severe fetal pathology and after legal authorization of medical termination of pregnancy given by the Multidisciplinary Center of Prenatal Diagnosis.

SUMMARY:
The aim of this study is to improve professional practices by better understanding parents who face the choice of medical termination of pregnancy.

The hypothesis of the study is that the decision to continue the pregnancy with a serious fetal pathology is more based on the belief and the representations of parents than on the diagnosis or prognosis criteria of the fetus.

A better understanding of the parents' motivations on their decision making by knowing what they expect from the caregivers would allow the division of representations, a better prenatal advice and a better perinatal support.

ELIGIBILITY:
Inclusion Criteria:

* Adults without age limit
* Couples or single mothers seen at hospital in 2019
* Couples or single mothers who have been taken care at the Antenatal Diagnosis Center
* Couples or single mothers whose file has been presented to a Multidisciplinary Prenatal Diagnosis Center (MPDC)
* MPDC's legal authorization of medical termination of pregnancy for severe fetal pathology (fetal reason)

Exclusion Criteria:

* MPDC's legal authorization of medical termination of pregnancy for maternal reason
* Parents who have requested an opinion on another MPDC (with continuation of care in another center)
* Fetal death in utero before couple's decision to continue or terminate the pregnancy
* Psychiatric pathology preceding the pregnancy
* Non-affiliation to health insurance plan
* No possible communication (language barrier)
* Participation refusal
* Adult patient protected under the terms of the law (Public Health Code)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be couples whose files were presented to the Multidisciplinary Prenatal Diagnosis Centers of two level 3 maternity hospitals in Lyon during 2019 for a severe fetal pathology, and for which the authorization of medical termination of pregnancy was delivered.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Quantitative auto-questionnaire (Likert scale) | 1 year
  Quantitative comparison of motivations related to the condition of the fetus versus motivations related to the beliefs and representations of the parents evaluated with a quantitative auto-questionnaire (Likert scale) completed more than one year after the diagnosis of severe fetal pathology.
  Each item of the questionnaire completed by parents who continued or terminated the pregnancy will be scored with a Likert scale. The sums of the Likert scores for the items concerning the fetus and the parental beliefs and representations will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie VIAUX-SAVELON, MD, Principal Investigator — Service d'obstétrique et de néonatologie, psychiatrie périnatale - Hôpital de la Croix-Rousse - Hospices Civils de Lyon
Locations (1):
- Service d'obstétrique et de néonatologie, psychiatrie périnatale - Hôpital de la Croix-Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided